CLINICAL TRIAL: NCT06687616
Title: Randomized Controlled Trial of Virtual Reality Therapies for Irritable Bowel Syndrome
Brief Title: RCT of VR Therapy for IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Almario (Other)
Collaborators: The Cleveland Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Christopher Almario, Associate Professor of Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY3343; R01DK140676 (NIH)
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: Virtual Reality; Cognitive Behavioral Therapy
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SynerGI (Experimental): The standardized CBT program (SynerGI) will be delivered through the Meta Quest 2 device and is self-administered and includes a network of environments arranged in a virtual clinic that participants experience at home though a protocolized, 8-week program. Depending on the module, experiences within the program last between 5-20 minutes. Participants will be prompted to regularly use the headset each week over the 8-week study period. The VR modules are reinforced with regularly scheduled messages and CBT exercises delivered by a webapp that is available on any smartphone or computer. The program progressively builds new skills and culminates in transitioning from using VR to applying the skills learned in VR to everyday life.
  Interventions: Device: SynerGI
- Sham VR (Sham Comparator): Patients in the sham VR group will receive the same Meta Quest 2 device but will only have access to a distraction-based VR therapy program that includes 2D nature videos (e.g., relaxing on a beach, swimming with dolphins). Similar to the SynerGI arm, people in the sham VR group will be prompted to regularly use the headset each week for the 8-week treatment period.
  Interventions: Device: Sham VR

INTERVENTIONS:
Device: SynerGI — Standardized 8-week CBT program, used for 20-30 minutes per week
  Arms: SynerGI
Device: Sham VR — Distraction-based VR program with 2D nature videos to be used for 8 weeks, 2-2 times a week for 10 minutes
  Arms: Sham VR

SUMMARY:
Through a pilot randomized controlled trial (RCT), the aim is to test the clinical impact and feasibility of a virtual reality (VR) cognitive behavioral therapy (CBT) program versus sham VR among patients with irritable bowel syndrome (IBS). It is hypothesized that using VR-administered CBT may reduce abdominal pain, leading to improved overall physical, psychological, and social functioning when compared to sham VR.

DETAILED DESCRIPTION:
A pilot randomized, sham-controlled clinical trial will be conducted in participants with IBS to achieve the following aims: Aim 1-collect preliminary data assessing the clinical impact of VR cognitive behavioral therapy (CBT) (SynerGI); Aim 2-establish the feasibility of using an 8-week VR CBT program among patients with IBS. The study will follow the established NIH protocol for conducting VR clinical trials, which aligns with VR-CORE clinical trial guidance. Participants will be randomized in a 1:1 ratio between two arms : (i) immersive VR CBT Program (SynerGI); and (ii) sham VR. As a pilot randomized controlled trial, it will not be powered for hypothesis testing of clinical outcomes . Instead, the focus will be on determining the plausibility and feasibility of SynerGI, with the aim to recruit 30 fully analyzable patients per arm.

Patients will be randomized 1:1 to each study arm . Block randomization will be implemented, using random permuted block sizes of 6, 8, or 10, allowing for up to 15% additional participants beyond the original sample size to account for dropouts. Randomization will also be stratified by sex to ensure a balance of women and men in each arm. Assessments will take place at baseline, midway through therapy at 4 weeks, and after completing the program at 8 weeks (a standard treatment length for VR trials).

ELIGIBILITY:
Inclusion Criteria:

* Has been diagnosed by a physician with Rome IV IBS; all subtypes will be included
* Has clinically significant abdominal pain as defined as an NIH PROMIS abdominal pain T-score ≥ 55 (0.5 standard deviation [SD] above the normalized population mean of 50)
* Able to read/write English (SynerGI is currently only available in English)
* Owns a compatible android or iOS smartphone, or personal laptop or desktop computer (excluding tablets) to complete surveys and has access to internet and email

Exclusion Criteria:

* Presents with a condition that interferes with VR usage, including history of seizure, facial injury precluding safe placement of headset, significant visual or hearing impairment that impacts ability to see the VR images or follow audio instructions
* Has cognitive impairment that would affect protocol participation
* Has a comorbid disorder that may confound the diagnosis of IBS, including celiac disease, inflammatory bowel disease, autoimmune disorders that affect the GI system, history of bowel resection, HIV/AIDS, diabetes with HgA1c >=7.0, neuroendocrine tumors, microscopic colitis, eosinophilic bowel disease, acute intermittent porphyria, or any other condition that a physician believes can mimic IBS symptoms and undermine diagnostic certitude
* Takes standing doses of opioid medications given the often severe impact of opioids on GI motility and potential for pharmacological visceral hyperalgesia
* Previously participated in a VR clinical trial
* Previously participated in talk therapy
* Previously used a VR program to treat their IBS

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
PROMIS Abdominal Pain Severity | Weekly; Baseline through Week 8
  Abdominal pain severity as measured by the 5-item PROMIS Abdominal Pain Severity scale. The scale is rendered using a T-statistic, where a score of 50 represents the population mean and 10 points is a SD.

SECONDARY OUTCOMES:
IBS-Symptom Severity Scale (IBS-SSS) | Baseline, Week 4 and Week 8
  IBS symptom severity as measured by the IBS-SSS. The maximum IBS-SSS score is 500, and patients can be categorized as having mild (75-175), moderate (176-300), and severe (>=300) symptoms.
IBS Quality of Life (IBS-QOL) | Baseline, Week 4 and Week 8
  IBS quality of life as measured by the IBS-QOL. The score range for the IBS-QOL is 0 to 100.

OTHER OUTCOMES:
Visceral Sensitivity Index (VSI) | Baseline, Week 4 and Week 8
  GI symptom-specific anxiety as measured by the VSI. The VSI is 15 items.
NIH PROMIS Depression | Baseline, Week 4 and Week 8
  Perceived depression as measured by the NIH PROMIS Depression scale. The scale is rendered using a T-statistic, where a score of 50 represents the population mean and 10 points is a SD.
NIH PROMIS Anxiety | Baseline, Week 4 and Week 8
  Perceived anxiety as measured by the NIH PROMIS Anxiety scale. The scale is rendered using a T-statistic, where a score of 50 represents the population mean and 10 points is a SD.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V Almario, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cleveland Clinic, Cleveland, Ohio

DOCUMENTS (1):
  • Informed Consent Form (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT06687616/ICF_000.pdf